CLINICAL TRIAL: NCT01565811
Title: Prospective Phase II Trial on Prophylactic Perihepatic Lymphadenectomy in Patients With Colorectal Cancer With Liver Metastasis
Acronym: LN
Status: Completed | Type: Observational
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Won-Suk Lee, Assistant Professor, Gachon University Gil Medical Center
Other Study IDs: girba2291
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Colorectal Cancer With Liver Metastasis
Keywords: colon neoplasm, rectal neoplasm, liver metastasis
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Hepatic pedicle lymph node Involvement: Intervention Type: perihepatic lymphadenectomy(surgical procedure)
  Interventions: Procedure: perihepatic lymphadenectomy

INTERVENTIONS:
Procedure: perihepatic lymphadenectomy — Hepatic pedicle lymph node dissection according to the protocol of the prospective multicentric study.Namely the six main groups of lymph nodes removed (HA,hepatic artery; CA, celiac axis; BD, common bile duct).

SUMMARY:
Objective: To evaluate the role of regional lymphadenectomy in patients with colorectal cancer liver metastasis. Background: Lymph node status is 1 of the most important prognostic factors in oncologic surgery; however, the role of lymph node dissection remains unclear for colorectal cancer liver metastasis.

DETAILED DESCRIPTION:
Lymph node status is a definite prognostic factor in oncologic surgery and significantly affects long-term survival, as reported by the tumor staging system of the International Union Against Cancer (IUCC), which is the most widespread classification of malignant tumors worldwide. Regional lymphadenectomy is already the standard procedure that completes hepatic resection in the case of carcinoma arising from the extrahepatic bile duct. However, the indication, extent, and role of lymph node excision are still a matter of discussion, and no clear guidelines exist in patients with colorectal cancer liver metastasis.

ELIGIBILITY:
Inclusion Criteria:

1. first hepatectomy;
2. age <75 years;
3. absence of severe cardiovascular,pulmonary, or other associated diseases;
4. absence of other malignant disease;
5. absence of distant metastases secondary to colorectal cancer other than liver metastases (except a solitary peritoneal tumor that could be completely resected during hepatectomy); and
6. complete resection of liver metastases confirmed during surgery.

Exclusion Criteria:

1. HNPCC
2. FAP
3. patient who refuses perihepatic lymphadnectomy
4. medical condition in which surgery cannot be tolerated

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Biopsy confirmed colorectal cancer with liver metastasis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-08; Primary Completion 2012-03 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
complication rate | within 3months

SECONDARY OUTCOMES:
To evaluate prognostic significance of perihepatic LN involvement with overall survival and disease free survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Won-Suk Lee, MD, Principal Investigator — Gil Hospital
Locations (1):
- Won-Suk Lee, Incheon, South Korea